CLINICAL TRIAL: NCT00033059
Title: Assessment of Potential Interactions Between Intravenous Cocaine and Tolcapone
Brief Title: Assessment of Potential Interactions Between Cocaine and Tolcapone - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0003-1; NCT00024765 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2003-08

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Tolcapone

INTERVENTIONS:
Drug: Tolcapone

SUMMARY:
The purpose of this study is to assess the potential interactions between intravenous (IV) cocaine and tolcapone.

DETAILED DESCRIPTION:
Double-blind, inpatient study by screening responses to cocaine infusions of 20 and 40 mg i.v. subjects into 1 of 2 treatment groups to assess potential interactions between i.v. cocaine infusion and treatment with tolcapone.

ELIGIBILITY:
Inclusion Criteria:

Volunteers dependent on cocaine and are non-treatment seeking; between 18-45 yrs of age; DSM-4 criteria for cocaine abuse or dependence

Exclusion Criteria:

Additional criteria available during screening at the site

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2001-07; Study Completion 2002-03

PRIMARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- UCLA Integrated Substance Abuse Program, Los Angeles, California, United States